CLINICAL TRIAL: NCT05508880
Title: SIGIL: Signal Interpretation and Analysis In Real Life Cardiac Arrhythmias
Acronym: SIGIL
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Heart Centre Singapore (Other)
Collaborators: Duke-NUS Graduate Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 2019/2774
Record Dates: First submitted 2022-08-18; First posted 2022-08-19 (Actual); Last update posted 2022-08-19 (Actual); Status verified 2022-08

CONDITIONS: Cardiac Arrhythmia
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study essentially consists of the prospective collection of mapping data derived from patients undergoing clinically indicated 3D mapping procedures. There is no intervention. The mapping data is used to construct and/or validate new activation mapping algorithms but will not be used to direct clinical treatment of the patient.

DETAILED DESCRIPTION:
Cardiac arrhythmias are a common clinical problem in cardiology. Often, such arrhythmias can be effectively and permanently treated through catheter ablation.

A key technology enabling the success of catheter ablation is activation mapping of cardiac arrhythmias. This refers to the construction of maps which depict the sequential activation of the cardiac chamber of interest. It is a fundamental electrophysiology technique, but at the same time, the principles behind activation map construction have not changed for decades.

In brief, the way activation maps are constructed nowadays consists of the following steps:

(i) Sequential acquisition of voltage signals throughout the cardiac chamber of interest, recording both the signal together with the location of the signal in 3D space (ii) Local activation time annotation of each of the acquired signals in relation to a so-called timing reference (iii) Depiction of the annotated activation time graphically as a so-called activation map, through which the mechanism of the arrhythmia can be understood and an appropriate ablation target chosen

Following assignment of the LAT to each individual signal, the map is complete and can be used to discern the arrhythmia circuit to choose an appropriate ablation target.

The objective of this study is to develop, refine and validate LAT-independent methods of activation map analysis using mapping data acquired from patients undergoing clinically indicated EP mapping and ablation procedures.

Specific objectives:

(i) Electrogram signature analysis. To use machine learning techniques to identify electrogram properties associated with specific conduction patterns.

(ii) Intracardiac EGM summation. To integrate all acquired points into a global function that allows as precise a determination as possible of the period of isthmus conduction in re-entrant arrhythmias.

(iii) Conduction velocity estimation. To algorithmically determine conduction velocity using proprietary techniques to wholly or partially reduce reliance on LAT annotation.This study aims to collect the electroanatomic 3D maps from patients to develop novel mapping algorithms, but this map data is not used to direct clinical treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patient undergoing a clinically indicated 3D mapping procedure for a cardiac arrhythmia
2. Ability to provide informed consent

Exclusion Criteria:

* Patients who cannot provide informed consent will be excluded. Otherwise, there are no specific exclusion criteria.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: At the National Heart Center Singapore, based on national audit data specific for NHCS, approximately 600 ablation procedures are performed per year, of which at least 150 would be expected to suitable for study inclusion. To recruit 40, we would only require ~25% participation rate which we think is realistic.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2019-10-30 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
The overall objective of this study is to develop, refine and validate LAT-independent methods of activation map analysis using mapping data acquired from patients undergoing clinicallyindicated EP mapping and ablation procedures. | 2 years
  This study aims to collect the electroanatomic 3D maps from patients to develop novel mapping algorithms, but this map data is not used to direct clinical treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart Centre Singapore, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No